CLINICAL TRIAL: NCT05509985
Title: A Phase 1 Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ASKG315 as a Single Agent and in Combination With Pembrolizumab in Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Study of ASKG315 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AskGene Pharma, Inc. (Industry)
Collaborators: Jiangsu Aosaikang Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASKG315-101
Record Dates: First submitted 2022-08-15; First posted 2022-08-22 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2022-08

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASKG315 (Experimental): Single or multiple ascending dose of ASKG315
  Interventions: Biological: ASKG315

INTERVENTIONS:
Biological: ASKG315 — Injection with dose escalation stage of 3mg up to 45mg as well as dose expansion stage with recommended dose level from dose escalation stage.

SUMMARY:
The study is a Phase 1, open-label, multicenter, dose escalation study to evaluate the safety, tolerability, PK and PD of ASKG315 as a single agent (Part 1) and in combination with pembrolizumab (Part 2) in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Each part of the study consists of 3 periods: screening (up to 28 days), treatment and follow-up. After an initial screening period, ASKG315 or ASKG315 combined with pembrolizumab will be administered once every 3 weeks by intravenous (IV) infusion. The Part 1 dose escalation consists of 6 planned escalation cohorts, with a starting dose of 3 mg. The Part 2 dose escalation consists of 4 planned escalation cohorts.

Part 2 of the study will begin enrolling after Part 1 has successfully and safely dosed all patients in the first two cohorts and followed these patients through the entire DLT period. The starting dose of Part 2 will be determined according to the safety and PK of ASKG315 in Part 1 of the study, but in no case will it exceed the highest dose already safely administered in Part 1 and confirmed as tolerable by the Safety Review Committee in Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Male or female ≥ 18 years of age (at the time signed consent is obtained).
3. Histologically or cytologically confirmed advanced malignant solid tumor that is refractory to or intolerant of all standard therapy or for which no standard therapy is available.
4. Measurable disease, per RECIST v1.1.
5. ECOG Performance Status of ≤ 2.
6. Life expectancy of ≥3 months, in the opinion of the Investigator.
7. Adequate organ function defined.
8. Fertile patients must be willing to use effective contraceptive measures (hormonal or barrier methods or abstinence, etc.) starting with the Screening visit through 90 days + 5 drug half-lives after the last dose of study treatment.
9. Negative serum pregnancy test for female patients within 7 days prior to the first dose of the study drug or documentation of lack of childbearing potential.
10. Willing and able to participate in the trial and comply with all trial requirements.

Exclusion Criteria:

Patients who meet any of the following criteria are not allowed to be enrolled:

1. Received any other investigational drug for treatment that is not commercially available within 4 weeks prior to Cycle 1 Day 1.
2. Received chemotherapy, radiotherapy, biotherapy, endocrine therapy, targeted therapy, immunotherapy, or any other anti-tumor treatments within 4 weeks prior to Cycle 1 Day 1.
3. Had major organ surgery or significant trauma within 4 weeks prior to C1D1 or planning elective surgery during the study period.
4. Received systemic glucocorticoid or other immunosuppressant treatment within 14 days prior to C1D1.
5. Received immunomodulatory drugs, including but not limited to thymosin and interferon, within 14 days prior to C1D1.
6. Received a live attenuated vaccine within 4 weeks prior to C1D1.
7. Received IL-2 or IL-15 therapy within 12 weeks prior to C1D1.
8. History of hematologic stem cell transplant or solid organ transplant.
9. Adverse reactions to previous antitumor therapy have not recovered to CTCAE 5.0 grade ≤ 1.
10. Cerebral parenchymal metastasis or meningeal metastasis with clinical symptoms.
11. Have an active infection that currently requires intravenous anti-infection therapy.
12. A history of human immunodeficiency virus (HIV) infection with a CD4+ T-cell count of ≤350 cells/µL at screening. HIV positive patients must be receiving adequate treatment.
13. If serological evidence of chronic hepatitis B virus infection (HBV), viral load below the limit of quantification at screening.
14. If serological evidence of hepatitis C virus infection (HCV), should have completed curative antiviral treatment and have HCV viral load below the limit of quantification at screening.
15. Current clinically significant interstitial lung disease.
16. History of serious cardiovascular or cerebrovascular diseases.
17. Active or recurrent autoimmune diseases.
18. History of Grade ≥ 3 Immune-Related Adverse Events (irAE) or Grade ≥ 2 immunotherapy-associated myocarditis associated with treatment with an immune checkpoint inhibitor.
19. Grade ≥ 3 bleeding .
20. Symptomatic with uncontrolled ascites or pleural effusion.
21. History of a grade ≥ 3 allergic reaction to protein drugs.
22. Known to have alcohol or drug dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-09 (Estimated); Primary Completion 2023-09-09 (Estimated); Study Completion 2024-09-09 (Estimated)

PRIMARY OUTCOMES:
Safety[DLTs、AEs、ECG] | 21days
  1. Incidence of dose limiting toxicities (DLTs)
  2. Incidence of adverse events (AEs), laboratory abnormalities, and ECG abnormalities

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 21days
  To evaluate the systemic pharmacokinetics of ASKG315 in subjects.
Area under the concentration time curve (AUC) | 21days
  To evaluate the systemic pharmacokinetics of ASKG315 in subjects.
Cytokine | 21days
  Changes in circulating cytokine levels.
Immunocyte | 21days
  Changes in immunocyte levels by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Hickingbottom, MD, Study Director — Ask-Gene Pharma, Inc.
Locations (2):
- Australia (2):
  - The Alfred Hospital, Melbourne
  - Blacktown Hospital, Sydney

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD or supporting information available.